CLINICAL TRIAL: NCT00195507
Title: A Randomized, Open Label Study to Evaluate the Safety and Efficacy of Etanercept in the Treatment of Subjects With Psoriasis
Brief Title: Study Evaluating Etanercept in the Treatment of Subjects With Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0881A6-101764
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2010-05-04 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2010-04

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
This study will provide a direct comparison of 'continuous therapy' and 'intermittent therapy' with withdrawal and retreatment upon return of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Stable, active plaque psoriasis
* Failure to respond to the following systemic therapies: Methotrexate, Cyclosporine, PUVA or Fumarate

Exclusion Criteria:

* Evidence of skin conditions other than psoriasis that would interfere with evaluations of the effect of the study
* Systemic psoriasis therapy within 28 days prior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2004-12; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Italy,Greece, decresg@wyeth.com; Trial Manager, Principal Investigator — For Denmark, Finland, Sweden, Norway, MedInfoNord@wyeth.com; TRial manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For Austria, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com; Trial Manager, Principal Investigator — For Hungary, WPBUMED@wyeth.com; Trial Manager, Principal Investigator — For Turkey, Erisc@wyeth.com; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For Germany, MedinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For UK, ukmedonfo@wyeth.com
Locations (114):
- Austria (2):
  - Feldkirch
  - Vienna
- Belgium (5):
  - Brussels
  - Edegem
  - Ghent
  - Leuven
  - Liège
- Prague, Czechia
- Denmark (3):
  - Aarhus C
  - Odense C
  - Roskilde
- Finland (2):
  - Kuopio
  - Lahti
- France (25):
  - Besançon
  - Bordeaux
  - Boulogne-Billancourt
  - Brest
  - Créteil
  - Dijon
  - Lille
  - Lyon
  - Marseille
  - Marseille Cédex 09
  - Montpellier Cédex 5
  - Nancy
  - Nantes
  - Nice
  - Nîmes
  - Paris
  - Pessac
  - Pierre-Bénite
  - Poitiers
  - Reims
  - Rouen
  - Saint-Etienne
  - Strasbourg
  - Toulouse
  - Tours
- Germany (15):
  - Bochum
  - Düsseldorf
  - Erlangen
  - Essen
  - Frankfurt
  - Hamburg
  - Kiel
  - Leipzig
  - Magdeburg
  - Mainz
  - Münster
  - Nordheide
  - Osnabrück
  - Tübingen
  - Würzburg
- Greece (2):
  - Athens
  - Thessaloniki
- Budapest, Hungary
- Italy (9):
  - Ancona
  - Cagliari
  - Genova
  - Modena
  - Padua
  - Pavia
  - Roma
  - Terni
  - Torino
- Netherlands (7):
  - Amsterdam
  - Capelle aan den IJssel
  - Heerlen
  - Nijmegen
  - Rotterdam
  - Utrecht
  - Voorburg
- Norway (3):
  - Bergen
  - Oslo
  - Stavanger
- Warsaw, Poland
- Lisbon, Portugal
- Spain (6):
  - Barcelona
  - Bilbao
  - Llobregat
  - Madrid
  - Málaga
  - Valencia
- Sweden (6):
  - Danderyds
  - Gothenburg
  - Linköping
  - Lund
  - Stockholm
  - Umeå
- Switzerland (3):
  - Basel
  - Bern
  - Geneva
- Turkey (Türkiye) (3):
  - Bornova-Izmir
  - Capa-Istanbul
  - Kocamustafapasa-Istanbul
- United Kingdom (19):
  - Aberdeen
  - Airdrie
  - Birmingham
  - Cardiff
  - Coventry
  - Dublin
  - Dundee
  - Glasgow
  - Lancaster
  - Leeds
  - Leicester
  - Liverpool
  - London
  - Newcastle upon Tyne
  - Newport
  - Norwich
  - Salford
  - Sheffield
  - Suffolk

REFERENCES:
- [Derived] Griffiths CE, Christophers E, Szumski A, Jones H, Mallbris L. Impact of early vs. late disease onset on treatment response to etanercept in patients with psoriasis. Br J Dermatol. 2015 Nov;173(5):1271-3. doi: 10.1111/bjd.13865. Epub 2015 Aug 17. No abstract available. PMID 25913550
- [Derived] Griffiths CE, Luger TA, Brault Y, Germain JM, Mallbris L. Retreatment in patients with psoriasis achieving response with etanercept after relapse due to treatment interruption: results from the CRYSTEL study. J Eur Acad Dermatol Venereol. 2015 Mar;29(3):468-73. doi: 10.1111/jdv.12585. Epub 2014 Aug 4. PMID 25087839

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in multiple countries worldwide from to.
Pre-assignment Details: Subjects were screened up to 4 weeks.
Groups:
- Continuous: etanercept 25 mg subcutaneously (SC) twice weekly for 54 weeks
- Intermittent: etanercept 50 mg SC twice weekly for 12 weeks, or less if a response was achieved earlier. If after 12 weeks there was an inadequate response or a relapse, etanercept 25 mg twice weekly was administered until a response was achieved.
Period: Overall Study
Arm/Group | Continuous | Intermittent
Started | 357 | 363
Completed | 258 | 245
Not Completed | 99 | 118
Not completed — Adverse Event | 24 | 13
Not completed — Death | 0 | 1
Not completed — Failed to Return | 4 | 3
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Protocol Violation | 5 | 4
Not completed — Lack of Efficacy | 40 | 67
Not completed — Withdrawal by Subject | 16 | 23
Not completed — Protocol Deviation | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous | Intermittent | Total
Number analyzed (Participants) | 357 | 363 | 720
Age Continuous [Mean (Standard Deviation); unit: years] | 44.87 (11.83) | 45.20 (11.88) | 45.03 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 102 | 203
  Male | 256 | 261 | 517
Region of Enrollment [Number; unit: participants]
  Portugal | 6 | 6 | 12
  Greece | 9 | 8 | 17
  Finland | 5 | 5 | 10
  Spain | 19 | 19 | 38
  Turkey | 7 | 11 | 18
  Austria | 13 | 11 | 24
  United Kingdom | 59 | 60 | 119
  Switzerland | 4 | 3 | 7
  Italy | 40 | 39 | 79
  France | 50 | 52 | 102
  Czech Republic | 3 | 3 | 6
  Hungary | 2 | 3 | 5
  Belgium | 22 | 21 | 43
  Poland | 5 | 5 | 10
  Denmark | 10 | 9 | 19
  Netherlands | 23 | 25 | 48
  Germany | 57 | 58 | 115
  Norway | 7 | 8 | 15
  Sweden | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Physician Global Assessment of Psoriasis (PGA) Score - Mean Value Over 54 Weeks
Description: Physician Global Assessment of Psoriasis (PGA) is a 7-point scale used to assess severity of psoriatic plaques (1=severe psoriasis, 7=clear).
Time Frame: 54 weeks
Population: The analysis population was the modified intention-to-treat (mITT)population, which included all patients who received at least one dose of study drug and had at least 1 post-baseline evaluation. Last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Continuous | Intermittent
Number analyzed (Participants) | 352 | 359
units on scale | 1.98 (0.86) | 2.51 (0.65)
Statistical Analysis 1: Comparison: Continuous vs Intermittent; Test type: Superiority or Other; p < 0.001, ANCOVA; Treatment and center as main effects, and baseline score as a covariant; Mean Difference (Net) = -0.53, 95% CI [-0.64 to -0.43]

2. Secondary Outcome: Patient Global Assessment of Psoriasis Score - Percentage of Improvement From Baseline
Description: Patients were asked to rate the severity of their psoriasis disease activity on a 6-point scale, where 0=good and 5=severe.
Time Frame: 54 weeks
Population: as for outcome 1
Measure: Number; unit: percentage improvement
Arm/Group | Continuous | Intermittent
Number analyzed (Participants) | 348 | 355
percentage improvement | 57.03 | 40.92
Statistical Analysis 1: Comparison: Continuous vs Intermittent; Test type: Superiority or Other; p < 0.001, ANCOVA

3. Secondary Outcome: Time to Achieve a Physician Global Assessment of Psoriasis Score of "Clear" or "Almost Clear"
Description: Physician Global Assessment of Psoriasis (PGA) is a 7-point scale used to assess severity of psoriatic plaques (1=sever psoriasis, 7=clear). This assessment measured the time (in days) from baseline to the visit where a patient achieved a PGA status of 0 or 1. Patients who did not achieve this status by their last visit were not included.
Time Frame: 54 weeks
Population: The analysis population was the modified intention-to-treat (mITT) population, which included all patients who received at least one dose of study drug, had at least 1 post-baseline evaluation and who achieved a PGA status of 0 or 1 by the last visit (Observed cases).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Continuous | Intermittent
Number analyzed (Participants) | 352 | 359
days | 127 [124 to 161] | 168 [126 to 253]

4. Secondary Outcome: Number of Patients With Survey Response of "Somewhat Satisfied" or Better
Description: Patients completed a patient satisfaction survey at baseline and throughout the study. Patients were asked to rate, based on their experienced during the past week, how satisfied or dissatisfied they were with their psoriasis therapy in general. Responses were based on a 7-point scale: Very satisfied, Satisfied, Somewhat Satisfied, Neutral, Somewhat Dissatisfied, Dissatisfied and Very Dissatisfied.
Time Frame: 54 weeks
Population: The analysis population was the modified intention-to-treat (mITT) population, which included all patients who received at least one dose of study drug and had at least 1 post-baseline evaluation.
Measure: Number; unit: participants
Arm/Group | Continuous | Intermittent
Number analyzed (Participants) | 352 | 359
participants
  Baseline | 70 | 80
  Week 54 | 231 | 198
Statistical Analysis 1: Comparison: Continuous vs Intermittent; Test type: Superiority or Other; p = 0.143, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Continuous | Intermittent
Serious Adverse Events (participants affected / at risk) | 23 | 31
Other Adverse Events (participants affected / at risk) | 281 | 273
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Continuous | Intermittent
Abdominal pain (General disorders) | 1/357 | 1/363
Abscess (General disorders) | 1/357 | 0/363
Accidental Injury (General disorders) | 3/357 | 2/363
Anaphylactoid reaction (General disorders) | 0/357 | 1/363
Back pain (General disorders) | 0/357 | 1/363
Cellulitis (General disorders) | 1/357 | 0/363
Hernia (General disorders) | 0/357 | 1/363
Infection (General disorders) | 1/357 | 2/363
Lab test abnormal (General disorders) | 1/357 | 0/363
Malaise (General disorders) | 1/357 | 0/363
Suicide attempt (Psychiatric disorders) | 0/357 | 1/363
Angina pectoris (Cardiac disorders) | 1/357 | 0/363
Cerebrovascular accident (Vascular disorders) | 0/357 | 1/363
Hypertension (Cardiac disorders) | 2/357 | 1/363
Left heart failure (Cardiac disorders) | 0/357 | 1/363
Myocardial infarct (Cardiac disorders) | 0/357 | 3/363
Myocardial ischemia (Cardiac disorders) | 1/357 | 0/363
Palpitation (Cardiac disorders) | 1/357 | 0/363
Varicose vein (Vascular disorders) | 1/357 | 0/363
Ventricular tachycardia (Cardiac disorders) | 0/357 | 1/363
Cholelithiasis (Hepatobiliary disorders) | 0/357 | 1/363
Gamma glutamyl transpeptidase increased (Hepatobiliary disorders) | 1/357 | 0/363
Gastroenteritis (Gastrointestinal disorders) | 1/357 | 0/363
Gastrointestinal carcinoma (Gastrointestinal disorders) | 0/357 | 1/363
Rectal disorder (Gastrointestinal disorders) | 1/357 | 0/363
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/357 | 1/363
Edema (Metabolism and nutrition disorders) | 1/357 | 0/363
Peripheral edema (Metabolism and nutrition disorders) | 1/357 | 0/363
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/357 | 0/363
Bone disorder (Musculoskeletal and connective tissue disorders) | 0/357 | 1/363
Synovitis (Musculoskeletal and connective tissue disorders) | 0/357 | 1/363
Ataxia (Nervous system disorders) | 1/357 | 0/363
Convulsion (Nervous system disorders) | 0/357 | 1/363
Dizziness (Nervous system disorders) | 1/357 | 0/363
Hypesthesia (Nervous system disorders) | 0/357 | 1/363
Incoordination (Nervous system disorders) | 0/357 | 1/363
Speech disorder (Nervous system disorders) | 0/357 | 1/363
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2/357 | 0/363
Nasal septum disorder (General disorders) | 1/357 | 0/363
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0/357 | 1/363
Erythema (Skin and subcutaneous tissue disorders) | 0/357 | 1/363
Psoriasis (Skin and subcutaneous tissue disorders) | 1/357 | 4/363
Skin carcinoma (Skin and subcutaneous tissue disorders) | 2/357 | 4/363
Abortion (Reproductive system and breast disorders) | 0/357 | 1/363
Kidney calculus (Renal and urinary disorders) | 1/357 | 0/363
Kidney pain (Renal and urinary disorders) | 1/357 | 0/363
Ovarian cyst (Reproductive system and breast disorders) | 0/357 | 1/363
Testis disorder (Renal and urinary disorders) | 1/357 | 0/363
Unintended pregnancy (Reproductive system and breast disorders) | 1/357 | 2/363
Urinary tract infection (Renal and urinary disorders) | 1/357 | 0/363
Urogenital disorder (Renal and urinary disorders) | 0/357 | 1/363
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Continuous | Intermittent
Accidental injury (General disorders) | 28/357 | 33/363
Asthenia (General disorders) | 27/357 | 22/363
Back pain (General disorders) | 26/357 | 18/363
Flu syndrome (General disorders) | 37/357 | 34/363
Headache (General disorders) | 63/357 | 47/363
Infection (General disorders) | 22/357 | 21/363
Injection site reaction (General disorders) | 21/357 | 24/363
Pain (General disorders) | 25/357 | 17/363
Hypertension (Cardiac disorders) | 19/357 | 10/363
Diarrhea (Gastrointestinal disorders) | 21/357 | 14/363
Metabolic and nutritional (Metabolism and nutrition disorders) | 19/357 | 23/363
Arthralgia (Musculoskeletal and connective tissue disorders) | 32/357 | 40/363
Nervous (Nervous system disorders) | 48/357 | 38/363
Cough increased (Respiratory, thoracic and mediastinal disorders) | 19/357 | 23/363
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 38/357 | 36/363
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 21/357 | 21/363
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 64/357 | 63/363
Pruritus (Skin and subcutaneous tissue disorders) | 33/357 | 28/363
Special senses (Ear and labyrinth disorders) | 29/357 | 20/363
Urogenital (Renal and urinary disorders) | 20/357 | 27/363

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.